CLINICAL TRIAL: NCT05681663
Title: The Effectiveness of Different Pressure of Extracorporeal Shock Wave Therapy for Management of Carpal Tunnel Syndrome: a Randomized Controlled Trial
Brief Title: The Effectiveness of Extracorporeal Shock Wave Therapy for Management of Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, İSMAİL CEYLAN, Dr., Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 43834581758
Record Dates: First submitted 2022-12-29; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.5 bar group (Experimental): 1. TENS, Parafin, exercise and In addition, 5 hertz 2000 pulses 1.5 bar ESWT will be applied to this group.
  Interventions: Other: Electroshock Wave therapy
- 4 bar group (Experimental): 1. TENS, Parafin, exercise and In addition, 5 hertz 2000 pulses 4 bar ESWT will be applied to this group.
  Interventions: Other: Electroshock Wave therapy

INTERVENTIONS:
Other: Electroshock Wave therapy — Randomized- Controlled trial
  Other Names: Parafin, Hotpack, Exercises, Splinting

SUMMARY:
Peripheral nerve entrapment neuropathies are the most common mononeuropathies in clinical practice. Carpal Tunnel Syndrome (CTS), n. It occurs as a result of compression of the medianus as it passes through the carpal tunnel, a narrow osteofibrous canal. CTS is the most common entrapment neuropathy of the upper extremity, affecting approximately 3% of the general adult population.

This study, which was designed as a randomized controlled study, will include 36 patients with CTS, aged between 18-65, who applied to Kırşehir Ahi Evran University Training and Research Hospital. In our study, both groups will be given 10 minutes of paraffin, 20 minutes of TENS, and 10 repetitions of tendon gliding exercise, 3 days a week for a total of 3 weeks (9 sessions). EESDT will be applied once a week in both groups (one group at 4 bar and the other at 1.5 bar pressure). Measurements will be made before treatment, after treatment, and at 12 weeks post-treatment.

In the literature, different pressure parameters were used in studies examining the efficacy of ESDT in the treatment of CTS. Although ESDT has been shown to have a curative effect on CTS, there is no consensus on which pressure parameter is more effective. Therefore, in this study, the effectiveness of ESDT applied at different pressure parameters in the treatment of CTS will be examined.

DETAILED DESCRIPTION:
Compression of peripheral nerves in fibroosseous tunnels located at segmental passages in the body is called entrapment neuropathy. In this type of neuropathies, the peripheral nerve is exposed to a neuropraxia-type injury in the area where it is compressed (1, 2). As a result, a picture develops in the distal part of the injured area, which leads to long-term motor, sensory and autonomic pathologies, and reduces the quality of life and functionality (3).

Carpal Tunnel Syndrome (CTS) occurs when the median nerve is exposed to compression during its passage through the carpal tunnel (4). Although CTS is the most common impingement neuropathy in the upper extremity, it has been reported to affect approximately 3% of the adult population (5). Although the incidence of CTS in women is three times higher than in men, the prevalence and severity increase with age. Work-related activities that require high-frequency repetition and force or the use of hand-operated vibrating tools significantly increase the risk of CTS (6).

CTS symptoms are generally characterized by pain and paresthesia in the innervation area of the median nerve in the hand region. Although these symptoms vary, they can sometimes be seen in the entire hand, rarely in the forearm and shoulder region. Repetitive wrist movements such as driving a vehicle, doing repetitive work with hand tools, squeezing diapers, and opening jars are activities that provoke the existing pathology. Patients generally report that their complaints decrease when they hold their hands down and shake them. This condition is known clinically as the Flick Sign and is 93% sensitive and 96% specific for CTS (7). As the anatomical localization within the carpal tunnel, the sensory fibers are subjected to compression before compared to the motor fibers, and only pain and paresthesia are seen in acute CTS. In severe cases where motor fibers are also affected, muscle weakness characterized by thumb abduction and oposition weakness is added to the present picture (8).

There are two different treatment options in CTS, conservative and surgical. In the conservative treatment of CTS; Conservative treatment methods such as local steroid injection, nonsteroidal anti-inflammatory drugs, diuretics, pyridoxine, splint, daily living activities, tendon-nerve slide exercises, manipulation, physical therapy, acupuncture, vitamin B6 are used. The approach in surgical treatment is surgical decompression and it is performed to relax the median nerve by loosening the transverse carpal ligament (9).

Eisenmenger defined the physical properties of extracorporeal shock wave therapy (ESDT) for the first time in 1959 and stated that high-intensity sound waves are applied to the body in the EIST treatment method (10). Shock waves were first applied to break up kidney stones in the 1980s. As the changes in the ilium were noticed while breaking the lower ureteral stones, studies were also started on bone tissues. Since 1990, research has been carried out on the use of this method in orthopedic diseases (11). ESDT has recently been widely used by orthopedists in Europe and the interest in its application has increased, and thousands of patients are treated with this method in the world (12).

Shock waves are caused by sudden changes in pressure, and these changes in pressure create strong waves that cause tension and compression. Shock wave is defined as acoustic wave. In sinusoidal shock waves, the pressure rises rapidly with a positive pressure (100-1000 bar) in as little as a few nanoseconds (ns) (less than 1 microsecond), followed by a rapid decrease and negative pressure.

The phase time of the wave is very short, the phase duration is defined in an average of 10 milliseconds (ms). Its frequency ranges from 16 hertz (Hz) to 20 megahertz (MHz). In this way, the energy is broken and reflected as it passes through areas such as bone and soft tissue, and the resulting kinetic energy affects the tissues. With the energy of the shock wave, cavitation occurs in the tissue and a force such as pressure and fragmentation occurs. Absorption of shock waves into the tissue is provided by conductive gels (11, 13).

In one study, a systematic review and analysis of randomized controlled trials was conducted on the effect of ESDT on CTS. In this study, 6 randomized controlled trials were examined. In conclusion, this meta-analysis revealed that ESDT can improve symptoms, functional outcomes and electrophysiological parameters in patients with CTS (10). In the literature, different pressure parameters have been used in studies examining the effectiveness of ESDT in the treatment of CTS (14,15,16). Although ESDT has been shown to have a curative effect on CTS (17), there is no consensus on which pressure parameter is more effective. Therefore, in this study, the effectiveness of ESDT applied at different pressure parameters in the treatment of CTS will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with Carpal Tunnel Syndrome

Exclusion Criteria:

* Those with systemic disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 6 week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir ahi Evran Üniversitesi, Kırşehir, Central Anatolia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceylan I, Kurtuncuoglu B, Tuncay F, Canli M, Alkan H, Tayfur A. Comparison of high- and low-dose radial extracorporeal shock wave therapy in carpal tunnel syndrome. Rev Assoc Med Bras (1992). 2025 May 2;71(3):e20241815. doi: 10.1590/1806-9282.20241815. eCollection 2025. PMID 40332277